CLINICAL TRIAL: NCT04351477
Title: The Effect of Mechanical Massage Chair on Musculoskeletal Pain Improvement for Endoscopists and Endoscopy Nurses
Brief Title: Mechanical Massage Chair on Musculoskeletal Pain Improvement
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Su Jin Chung, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 20200413
Record Dates: First submitted 2020-04-14; First posted 2020-04-17 (Actual); Last update posted 2020-04-22 (Actual); Status verified 2020-04

CONDITIONS: Massage Therapy
Keywords: massage chair; mulsculoskeletal pain

STUDY DESIGN:
Intervention Model Description: Randomized, open-label, cross-over study
Masking Description: 1. Randomization by allocation concealment
  2. Open label, cross-over design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Massage chair group (Experimental): Use mechanical massage chair for 20 minutes/1 session, 3 sessions/week, for 3 weeks
  Interventions: Device: Massage chair
- Control (No Intervention): No use of mechanical massage chair for 3 weeks

INTERVENTIONS:
Device: Massage chair — Mechanical massage chair
  Other Names: Bodyfriend
  Arms: Massage chair group

SUMMARY:
The effect of mechanical massage chair on musculoskeletal pain improvement for endoscopists and endoscopy nurses

DETAILED DESCRIPTION:
Randomized, open-label, cross-over study

1. 1st phase Massage chair group (20 minutes/session, 3 sessions/week, 3 weeks), vs. control (no use of massage chair)
2. Wash-out period (9 weeks)
3. 2nd phase (cross-over) Massage chair group (20 minutes/session, 3 sessions/week, 3 weeks), vs. control (no use of massage chair)

   * Msculoskeletal pain questionnaires (VAS, NDI, SPADI)

1) 1st phase: at baseline, 1.5 wk, 3 wk 2) 2nd phase: at baseline, 1.5 wk, 3 wk, 9wk after the end of treatment

ELIGIBILITY:
Inclusion Criteria:

* Endoscopists or endoscopic nurses working at Seoul National University Hospital Gangnam Center

Exclusion Criteria:

* Spine disease, skin disease, acute inflammation, electrical heart device, thromboembolism, fracture, osteoporosis, varicose vein
* Pregnancy

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2020-06-01 (Estimated); Primary Completion 2021-04-30 (Estimated); Study Completion 2021-04-30 (Estimated)

PRIMARY OUTCOMES:
Visual analogue scale | The change of VAS value at baseline, 1.5 week, 3 weeks during treatment, and 9 weeks after treatment
  range: 0-10 (0: no pain; 10: worst possible pain)

SECONDARY OUTCOMES:
Neck disability index (NDI) | The change at baseline, 1.5 week, 3 weeks during treatment, and 9 weeks after treatment
  range: 0-50 score (0: no pain or no disability, 50: worst pain or disability)
Shoulder pain and disability index (SPADI) | The change at baseline, 1.5 week, 3 weeks during treatment, and 9 weeks after treatment
  range: 0-100% (0: no pain or no disability, 100: worst pain or disability)

CONTACTS AND LOCATIONS:
Overall Officials: Min-Sun Kwak, MD, PhD, Principal Investigator — Seoul National University Hospital Gangnam Center
Locations (1):
- Healthcare System Gangnam Center, Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No